CLINICAL TRIAL: NCT07386665
Title: Impact of Circadian Exercise on Metabolic Dysfunction-Associated Steatotic Liver Disease in Postmenopausal Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Juan Manuel Alcantara Alcantara, Investigador Ramón y Cajal, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UALBIO2025/008
Record Dates: First submitted 2025-09-16; First posted 2026-02-04 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease; Cardiometabolic Diseases; Exercise
Keywords: Exercise; Metabolism; Health; Women
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual-Care Control Group (Placebo Comparator)
  Interventions: Behavioral: Usual-care control group
- Morning Exercise Group (Experimental)
  Interventions: Behavioral: Morning exercise group
- Evening Exercise Group (Experimental)
  Interventions: Behavioral: Evening exercise group

INTERVENTIONS:
Behavioral: Morning exercise group — Participants perform supervised exercise sessions at 07:00h
  Arms: Morning Exercise Group
Behavioral: Evening exercise group — Participants perform supervised exercise sessions at 19:00h
  Arms: Evening Exercise Group
Behavioral: Usual-care control group — Participants receive lifestyle counseling without exercise
  Arms: Usual-Care Control Group

SUMMARY:
Type of Study: Clinical Trial

Goal: The goal of this clinical trial is to investigate how performing exercise at different times of day (morning vs. evening) affects liver fat, cardiometabolic health, and gut microbiota in postmenopausal women.

Participant Population/Health Conditions: The study will involve 63 sedentary postmenopausal women (aged 45-75) diagnosed with metabolic dysfunction-associated steatotic liver disease.

Main Questions: The main questions this study aims to answer are:

* Does morning exercise reduce hepatic fat more effectively than evening exercise?
* How does time-of-day-specific exercise influence cardiometabolic markers?
* Do changes in gut microbiota contribute to the metabolic effects of exercise timing?

Participants Will:

Be randomized into one of three groups: morning exercise, evening exercise, or a usual-care control group.

Follow the assigned regimen for 12 weeks. The exercise groups will perform supervised aerobic and resistance training three times per week.

Provide blood, stool, and imaging data before and after the intervention to determine the effects of the intervention.

Comparison Group:

Researchers will compare the effects of morning vs. evening exercise (and usual care) on hepatic fat reduction and cardiometabolic improvement, as well as changes in gut microbiota.

DETAILED DESCRIPTION:
Metabolic dysfunction-associated steatotic liver disease (MASLD) affects approximately one in three adults and is a major contributor to the growing burden of cardiometabolic disease. Exercise is one of the most effective interventions for improving cardiometabolic health, reducing hepatic fat, and enhancing metabolic flexibility. However, the timing of exercise -a modifiable behavioral factor- may play a crucial yet underexplored role in determining its physiological benefits.

Preclinical studies have shown that circadian rhythms regulate key metabolic processes, including lipid metabolism and glucose homeostasis. Moreover, recent findings suggest that exercise performed at different times of day may elicit different responses, influencing the regulation of hepatic fat and systemic inflammation. These effects may be mediated, in part, through gut microbiota, which modulate host metabolism via the gut-liver axis. However, the interaction between exercise timing and gut microbiota in human physiology -particularly in women- remains poorly understood.

This knowledge gap is particularly critical in postmenopausal women, a population that experiences profound metabolic changes due to hormonal decline, including increased hepatic and visceral fat, chronic inflammation, and reduced insulin sensitivity. These alterations significantly elevate the risk for MASLD and other cardiometabolic diseases. Yet, postmenopausal women are consistently underrepresented in clinical trials exploring exercise interventions.

Based on emerging scientific evidence, the investigators hypothesize that morning exercise may lead to greater reductions in hepatic fat and improvements in cardiometabolic health compared to evening exercise in postmenopausal women with MASLD. Furthermore, the investigators propose that these effects may be partially mediated by exercise-induced changes in gut microbiota composition and function.

Thus, the main objective of the project is to investigate whether the timing of exercise modulates hepatic fat reduction, cardiometabolic adaptation, and gut microbiota remodeling in postmenopausal women with MASLD. To achieve this, the project will implement a randomized controlled trial in which 63 sedentary postmenopausal women diagnosed with MASLD will be randomly allocated into one of three groups: (i) morning exercise (07:00h), (ii) evening exercise (19:00h), or (iii) a usual-care control group receiving lifestyle counseling.

Participants in the intervention groups will complete a 12-week supervised training program, combining aerobic and resistance exercise (3 sessions/week, 60-90 minutes per session), in accordance with WHO recommendations. Before and after the intervention, biological samples, magnetic resonance imaging, and metabolic assessments will be collected. The study will employ advanced multi-omics analyses, including metabolomics and semi-targeted metagenomics, to explore how gut microbiota changes relate to improvements in metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 45-75 years, postmenopausal for at least two years (stage +1a)
* Body Mass Index (BMI) > 25 and < 40 kg/m²
* Diagnosed hepatic steatosis (via ultrasound hyperechogenicity, FibroScan CAP score >280, or histological confirmation)
* Sedentary lifestyle (no regular structured exercise)
* Willingness to be randomized and adhere to study procedures, including all assessments and visits
* Sufficient Spanish proficiency to understand and follow study instructions
* Consent to store biological samples for future research

Exclusion Criteria:

* Contraindications for MRI (e.g., claustrophobia, pacemaker, metal implants)
* History of major cardiovascular, endocrine, neurological, or kidney disease, or any clinical abnormalities (to be judged by the study physician)
* First-degree family history of sudden cardiac death
* Alcohol or substance abuse
* Psychiatric, psychotic, eating, or sleep disorders (to be judged by the study physician)
* Prior bariatric surgery, diagnosed HIV/AIDS, or inflammatory/autoimmune diseases
* Cancer or any medical condition where exercise is contraindicated (to be judged by the study physician)
* Recent or unstable metabolic conditions (e.g., diabetes, recent medication changes, or use of drugs affecting metabolism)
* Recent (<3 months) use of antibiotics, statins, glucocorticoids, hormonal therapies, amiodarone, or myelosuppressive agents
* Participation in weight-loss programs or special diets (e.g., ketogenic, high-carb)
* Shift workers or caregivers with frequent nocturnal disruptions

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 63 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Hepatic fat content | Change from baseline in the mean adipose tissue content at 12 weeks
  Hepatic fat content will be quantified using MRI

SECONDARY OUTCOMES:
Visceral adipose tissue | Change from baseline in the mean adipose tissue content at 12 weeks
  Visceral adipose tissue will be quantified using MRI
Intra-muscular adipose tissue | Change from baseline in the mean adipose tissue content at 12 weeks
  Intra-muscular adipose tissue, at the mid thigh, will be quantified using MRI
Body composition | Change from baseline in the whole-body composition at 12 weeks
  Whole-body composition will be quantified using DXA. Fat mass (in kg), and lean mass (in kg) will be assessed
Bone related parameters | Change from baseline in the whole-body mineral density and content at 12 weeks
  Whole-body bone related parameters will be quantified using DXA. Bone mineral density and content (both in g/cm^2) will be assessed
Resting blood pressure | Change from baseline in the resting blood pressure related parameters at 12 weeks
  Systolic pressure (mmHg) and diastolic pressure (mmHg) will be measured.
Glucose metabolism | Change from baseline in the glucose related parameters at 12 weeks
  Glucose metabolism (mg/dl) will be assessed via an oral glucose tolerance test with serial glucose measurements. Continuous glucose monitoring systems will be used to monitor 24-hour glycemic fluctuations (mg/dl) under free-living conditions
Energy metabolism | Change from baseline in the energy metabolism related parameters at 12 weeks
  Resting energy expenditure and exchange ratio will be determined using indirect calorimetry. Exercise energy expenditure and exchange ratio will be assessed during a steady-state submaximal exercise at 40-60% of VO2max
Exercise performance | Change from baseline in the exercise performance related parameters at 12 weeks
  VO2max will be assessed following an incremental test to exhaustion. Muscular strength will be evaluated through 1-RM for both upper and lower body muscular strength
Heart rate and heart rate variability | Change from baseline in the heart rate and heart rate variability related parameters at 12 weeks
  Heart rate (maximum and minimum values) and heart rate variability will be assessed at both, rest and exercise periods
Body weight | Change from baseline in the body weight at 12 weeks
  Body weight (in kg) will be assessed using a scale.
Height | Change from baseline in the height at 12 weeks
  Height (in m) will be assessed using a stadiometer.
Body mass index | Change from baseline in the height at 12 weeks
  Body weight (in kg) and height (in m) will be combined to report BMI in kg/m^2
Fasting glucose levels | Change from baseline in the fasting glucose levels at 12 weeks
  Fasting blood samples will be analyzed to determine glucose levels (mg/dl).
Fasting insulin levels | Change from baseline in the fasting insulin levels at 12 weeks
  Fasting blood samples will be analyzed to determine insulin levels (µmol/L).
Fasting HbA1c levels | Change from baseline in the fasting HbA1c levels at 12 weeks
  Fasting blood samples will be analyzed to determine HbA1c levels (mmol/mol).
Fasting cholesterol, high-density lipoprotein (HDL), and low-density lipoprotein (LDL) levels | Change from baseline in the fasting cholesterol, HDL, and LDL levels at 12 weeks
  Fasting blood samples will be analyzed to determine cholesterol, HDL, and LDL levels (mg/dl).
International Physical Activity Questionnaire | Change from baseline in the questionnaire score at 12 weeks
  The International Physical Activity Questionnaire (IPAQ) will be used for quantifying total physical activity in Metabolic Equivalent of Task-minutes per week (MET-min/week). In this questionnaire, a higher score indicates a greater volume of physical activity
Morningness-Eveningness Questionnaire | Change from baseline in the questionnaire score at 12 weeks
  The Morningness-Eveningness Questionnaire (MEQ) will be used for determining the individual's circadian typology. In this questionnaire, a higher score indicates a stronger "morning-type" preference and a lower score signifies an "evening-type" preference
Pittsburgh Sleep Quality Index Questionnaire | Change from baseline in the questionnaire score at 12 weeks
  The Pittsburgh Sleep Quality Index (PSQI) will be used for assessing subjective sleep quality and disturbances over a one-month period. In this questionnaire, a higher score represents poorer sleep quality; a score exceeding 5 typically denotes clinically poor global sleep
Three-Factor Eating Questionnaire | Change from baseline in the questionnaire score at 12 weeks
  The Three-Factor Eating Questionnaire (TFEQ) or TFEQ-R18 will be used for measuring three components of eating behavior (Cognitive Restraint, Emotional Eating, and Uncontrolled Eating). In this questionnaire, elevated subscale scores indicate more disordered or problematic eating patterns
Perceived Stress Scale Questionnaire | Change from baseline in the questionnaire score at 12 weeks
  The Perceived Stress Scale (PSS) will be used for measuring the degree to which life situations are appraised as stressful. In this questionnaire, a higher total score indicates a higher level of perceived psychological stress
Depression, Anxiety, and Stress Scale Questionnaire | Change from baseline in the questionnaire score at 12 weeks
  The Depression, Anxiety, and Stress Scale (DASS-21) will be used for providing three independent severity subscales (Depression, Anxiety, and Stress). In this questionnaire, an increased score on any subscale signifies a greater severity of symptomatology and a diminished mental health status
Beck Depression Inventory Questionnaire | Change from baseline in the questionnaire score at 12 weeks
  The Beck Depression Inventory (BDI-II) will be used for measuring depressive symptom severity. In this questionnaire, a higher score correlates directly with greater depressive symptom severity
Profile of Mood States Questionnaire | Change from baseline in the questionnaire score at 12 weeks
  The Profile of Mood States (POMS) will be used for assessing transient mood states. In this questionnaire, higher scores on negative subscales indicate a poorer mood state, while an increased score on the Vigor scale indicates a more favorable mood

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Almería, Almería, Spain